CLINICAL TRIAL: NCT00440284
Title: Flexible, Intensive vs. Conventional Insulin Therapy in Insulin-Naive Adults With Type 2 Diabetes - a Non-Blinded, Randomized Controlled Cross-Over Clinical Trial of Metabolic Control and Patient Preference
Brief Title: Flexible, Intensive vs. Conventional Insulin Therapy in Insulin-Naive Adults With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Jena (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1b
Record Dates: First submitted 2007-02-21; First posted 2007-02-27 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Type 2 Diabetes
Keywords: conventional insulin therapy; intensive insulin therapy; self-management; patient education; RCT; glycosylated hemoglobin; hypoglycemia; patient preference
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: conventional vs. flexible, intensive insulin therapy

SUMMARY:
Objective. Flexible, intensive insulin therapy (FIT) with pre-prandial regular insulin and conventional insulin therapy (CIT) with twice daily premixed insulin are treatment options in patients with type 2 diabetes who become insulin dependent. While intensive insulin therapy can increase meal and life style flexibility, conventional therapy is easier to perform. The aim of the study was to compare metabolic outcomes and patient preferences of both treatment regimens.

Research Design and Methods. Non-blinded, randomized controlled cross-over clinical pilot trial. Insulin naive participants who failed therapeutic goals under oral antidiabetic therapy underwent FIT and CIT for two months. Patients completed standard Diabetes Treatment and Teaching Programs (DTTP) and trained FIT and CIT. Main outcome measures were glycosylated hemoglobin (GHb), mild and severe hypoglycemia, insulin dosage, blood pressure and body-mass-index (BMI). Before/after and inter-group analyses were performed. Finally, therapy preference was analyzed.

DETAILED DESCRIPTION:
Hypothesis In the undertaken study we tested the hypothesis that flexible, intensive and conventional insulin therapy in insulin-naive adults with type 2 diabetes are equally effective in regards to metabolic outcomes. We hypothesized that younger participants in employment would prefer flexible, intensive insulin therapy.

Flexible, intensive and conventional insulin therapy CIT consisted of twice daily injections of premixed insulin (30% regular insulin, 70% NPH-insulin) before breakfast and dinner. Participants followed individually adjusted diet plans with fixed amounts of carbohydrates. Daily blood-glucose self-control was performed before insulin injections. Participants documented blood glucose readings and insulin dosage. Limited self-adjustment of insulin dosage was taught and encouraged in the DTTP, i.e. variance of up to 4 IU insulin per injection.

In FIT, participants measured blood glucose before main meals and at bedtime and adjusted regular insulin dosages to actual blood glucose levels and their desired carbohydrate intake on a meal by meal basis. When necessary, NPH insulin was added at bedtime. Additional administration of oral antidiabetic drugs was not permitted.

Study design, randomization and intervention The trial was designed as a clinical, prospective, randomized, non-blinded, single center, cross-over pilot study.

After randomization, participants started insulin therapy either with FIT or CIT and completed a Diabetes Treatment and Teaching Program on an out-patient basis. In this four week run-in period with weekly visits, individual insulin dosage and carbohydrate intake was determined (figure 1). The run-in was followed by an 8 week study sequence until cross-over. At cross-over, participants were given one structured teaching session for refreshing and switched from CIT to FIT (Group A) or FIT to CIT (Group B), respectively. After a one week run-in period for insulin dose-adjustment, participants completed the second 8 week study sequence. Regular visits were held at the beginning and at the end of both study sequences. Additional visits were held after 2 weeks, to adjust therapy if necessary. During visits, a study team consisting of a diabetologist and a specially trained nurse educator analyzed personal diabetes records and gave advice regarding insulin dose adjustment and other problems related to current diabetes therapy. At the end of the trial, participants decided which therapy to continue.

Setting, eligibility criteria and outcome measures Participants were recruited in the outpatient clinic of the Unit of Endocrinology and Metabolic Diseases of the Department of Internal Medicine of the Friedrich-Schiller-University, Jena.

All patients with type 2 diabetes who failed to achieve their therapeutic goals under oral antidiabetic therapy and who were referred by local General Practitioners to the outpatient clinic for initiation of insulin therapy were candidates for inclusion in the study. Participants who agreed to participate in the study were recruited in consecutive order as they were referred to the out-patient clinic. They were not admitted to the study if any of the following criteria were present: (1) not type 2 diabetes, (2) diabetes duration <2 years, (3) not insulin naive, (4) ineffective oral antidiabetic therapy < 3 months, (5) GHb below 7 or above 11%, (6) age below 40 or above 65 years, (7) co-medication with corticosteroids, (8) pregnancy, severe mental or somatic diseases or (9) unwillingness to return for follow-up.

The primary end-point with respect to the effectiveness of FIT and CIT was glycosylated (GHb). Secondary end-points were mild and severe symptoms of hypoglycemia, insulin dosage, blood pressure, BMI and individual therapy preference.

Sample size To have a 90% chance of detecting as significant (at the two sided 5% level) a 0.5 % difference between the two groups in GHb, with an assumed standard deviation of 0.8%, 38 participants were required.

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 2 diabetes who failed to achieve their therapeutic goals under oral antidiabetic therapy and who were referred by local General Practitioners to the outpatient clinic for initiation of insulin therapy were candidates for inclusion in the study.
* Participants who agreed to participate in the study were recruited in consecutive order as they were referred to the out-patient clinic.

Exclusion Criteria:

* Not type 2 diabetes,
* Diabetes duration <2 years,
* Not insulin naive,
* Ineffective oral antidiabetic therapy < 3 months,
* GHb below 7 or above 11%,
* Age below 40 or above 65 years,
* Co-medication with corticosteroids,
* Pregnancy, severe mental or somatic diseases or
* Unwillingness to return for follow-up.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2004-01; Study Completion 2004-12

PRIMARY OUTCOMES:
glycosylated hemoglobin (GHb)

SECONDARY OUTCOMES:
mild and severe hypoglycemia, insulin dosage, blood pressure and body-mass-index (BMI).

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kloos, MD, Principal Investigator — Klinik Innere Medizin III, Medical School, Friedrich Schiller University
Locations (1):
- Medical School, Friedrich Schiller University Jena, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Kloos C, Samann A, Lehmann T, Braun A, Heckmann B, Muller UA. Flexible intensive versus conventional insulin therapy in insulin-naive adults with type 2 diabetes: an open-label, randomized, controlled, crossover clinical trial of metabolic control and patient preference. Diabetes Care. 2007 Dec;30(12):3031-2. doi: 10.2337/dc07-0397. Epub 2007 Aug 23. No abstract available. PMID 17717285